CLINICAL TRIAL: NCT02022891
Title: The Impact of Systematic Psychological and Medical Care for Treatment of Pediatric Patients With SCD: : A Luxury or a Necessity?
Brief Title: Systematic Psychological and Medical Care for Children With SCD
Acronym: Drépano
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SC_MOE_2012-6
Record Dates: First submitted 2013-08-28; First posted 2013-12-30 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle cell disease; psychological support; quality of life
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- systematic psychological care: Systematic psychological treatment plan added to medical care for children with SCD. Bio-psychosocial paradigm applied at pediatric consultations.
- Control: medical care only at routine pediatric consultations for SCD. Psychological support provided only when the pediatrician consider it appropriate.
  Interventions: Behavioral: systematic psychological care

INTERVENTIONS:
Behavioral: systematic psychological care — Prevention treatment plan that provides systematic medical and psychological care at routine pediatric consultations for SCD. Bio-psychosocial paradigm applied at pediatric consultations.
  Groups: Control

SUMMARY:
Sickle cell disease (SCD), a genetically transmitted blood disease, necessitates life-long care. In children, the disease may cause intense pain and other severe complications. Studies show that sources of stress, as well as complex psychological and intercultural issues associated with SCD, often aggravate symptoms. At Louis Mourier hospital, the treatment model used is systematic psychological and medical care. Our hypothesis is that this care is beneficial for both the children and their families as seen in improved quality of life and positive impact on medical symptoms.

DETAILED DESCRIPTION:
In this observational multicentric pilot study, our goal is to assess the effectiveness of a systematic medical-psychological approach in place for the past 6 years at the Louis Mourier Hospital, as compared to the usual practice in 2 other pediatric hospitals for SCD which focus essentially on the medical issues associated with SCD. Two psychologists will interview 80 children and their primary care-takers at Louis Mourier hospital, and 80 children and their care-takers of the other two centers, using a standard comprehensive care for SCD. For the parents, we propose to use a semi-structured interview including a prepared interview guide, the Loneliness Questionnaire, and the parents' version of KIDSCREEN (10 items). For the children, according to their age, The Rey-Osterrieth Complex Figure Test (ROCF), the Draw a Person in the Rain Test (DPR), the KIDSCREEN questionnaire, and semi-directed interview will be used. Relevant information from the patients' medical record directly related to the symptomatic expression of the SCD will be noted on a data collection form. This phase is scheduled to last 12 months. A statistical and qualitative analysis of the results will be carried out at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* children with sickle cell disease
* treated in one of the three investigational centers
* All major forms of the disease will be studied regardless of the country of origin.

Exclusion Criteria:

* Refusal of the parents or the child to participate.
* Child or parent living in France for less than 6 months

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with sickle cell disease
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
psychological assessment and quality of life (quantitative and qualitative assessment) | baseline
  quality of life (scales, semi-directive interviews, drawings), psychological assessment of the children and their parent

SECONDARY OUTCOMES:
use of care-facilities: comparison between groups | baseline
  retrospective (back to 2006) collection of the number of hospitalizations (with mean length of stay) and number of emergency care experiences (and reasons) , number of children requiring the support of other care professionals for their SCD (Medico-Psychological center, orthophonist, neuro-pediatrician, psychologist..)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène ODIEVRE, MD, Principal Investigator — Hôpital Louis Mourier, Colombes, France 92
Locations (1):
- Hôpital Louis Mourier, Colombes, France